CLINICAL TRIAL: NCT05999825
Title: Safety and Preliminary Efficacy of Sm-p80 + GLA-SE (SchistoShield®) Vaccine Against Controlled Human Schistosome Infection in Healthy, Schistosoma-naïve Adults
Brief Title: Sm-p80 Schistosomiasis Challenge Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Leiden University Medical Center (Other)
Collaborators: Texas Tech University Health Sciences Center (Other); MRC/UVRI and LSHTM Uganda Research Unit (Other)
Responsible Party: Principal Investigator, Meta Roestenberg, Prof., Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Sm-p80
Record Dates: First submitted 2023-08-11; First posted 2023-08-21 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Schistosoma Mansoni; Schistosomiasis
MeSH Terms: conditions — Schistosomiasis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Vaccine group (Experimental): The vaccine group will be immunised three times with 30 μg Sm-p80 + 5 μg GLA-SE i.m. at weeks 0,4, and 8. Participants will be exposed to 20 male Schistosoma mansoni cercariae at week 12.
  Interventions: Biological: Sm-p80 + GLA-SE Vaccine; Biological: Schistosoma mansoni infection
- Placebo control group (Placebo Comparator): The placebo control group will be immunised three times with saline i.m. at weeks 0,4, and 8. Participants will be exposed to 20 male Schistosoma mansoni cercariae at week 12.
  Interventions: Other: Placebo; Biological: Schistosoma mansoni infection

INTERVENTIONS:
Biological: Sm-p80 + GLA-SE Vaccine — 30 μg Sm-p80 + 5 μg GLA-SE
  Arms: Vaccine group
Other: Placebo — 0.9% Sterile Normal Saline
  Arms: Placebo control group
Biological: Schistosoma mansoni infection — 20 viable male Schistosoma mansoni cercariae of the Puerto Rican strain

SUMMARY:
The goal of this clinical trial is to learn about the Sm-p80 + GLA-SE (Schistoshield®) vaccine in healthy participants who have not had schistosomiasis before. The main questions it aims to answer are:

* if the vaccine is safe
* if after vaccinated people start producing antibodies
* if the vaccine works against schistosomiasis.

Participants will receive three vaccines (or placebo) and are then exposed to 20 male Schistosoma cercariae. Afterwards they are treated with praziquantel to cure the infection.

Researchers will compare the group vaccinated with Schistoshield® and placebo (fake vaccination) to see if the vaccine has worked.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is aged ≥ 18 and ≤ 45 years and in good health.
2. Subject has adequate understanding of the procedures of the study and agrees to abide strictly thereby.
3. Subject is able to communicate well with the investigator, is available to attend all study visits.
4. Subject will not travel to Schistosoma-endemic countries up until treatment at week 24.
5. Subject agrees to refrain from blood and plasma donation to Sanquin or for other purposes throughout the study period.
6. For female subjects: subject agrees to use adequate contraception and not to breastfeed for the duration of study.
7. Subject has signed informed consent.

Exclusion Criteria:

1. Any history, or evidence at screening, of clinically significant symptoms, physical signs or abnormal laboratory values suggestive of systemic conditions, such as cardiovascular, pulmonary, renal, hepatic, neurological, dermatological, endocrine, malignant, haematological, infectious, immune-deficient, (severe) psychiatric and other disorders, which could compromise the health of the participant during the study or interfere with the interpretation of the study results. These include, but are not limited to, any of the following:

   * body weight <50 kg or Body Mass Index (BMI) <18.0 or >35.0 kg/m2 at screening;
   * positive HIV, HBV or HCV screening tests;
   * the use of immune modifying drugs within three months prior to study onset (inhaled and topical corticosteroids and oral anti-histamines exempted) or expected use of such during the study period;
   * history of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years;
   * any history of treatment for severe psychiatric disease by a psychiatrist in the past year;
   * history of drug or alcohol abuse interfering with normal social function in the period of one year prior to study onset.
2. The chronic use of any drug known to interact with praziquantel, artesunate or lumefantrine metabolism (e.g. phenytoïn, carbamazepine, phenobarbital, primidon, dexamethason, rifampicine, cimetidine, flecaïnide, metoprolol, imipramine, amitriptyline, clomipramine, class IA and III anti-arrythmics, antipsychotics, antidepressants, macrolides, fluorchinolones, imidazole- and triazole antimycotics, antihistamines). Because lumefantrine may cause extension of QT-time, chronic use of drugs with effect on QT interval will result in exclusion from study participation.
3. Any planned vaccination within 28 days before the start of the trial until the end of the immunisation phase (week 12), with the exception of SARS-CoV-2 vaccines or influenza vaccines.
4. For female subjects: positive serum pregnancy test on the day before first immunisation.
5. Any history of schistosomiasis or treatment for schistosomiasis.
6. Positive serology for schistosomiasis or elevated serum CAA at screening.
7. Known hypersensitivity to or contra-indications (including co-medication) for use of praziquantel, artesunate or lumefantrine.
8. Being an employee or student of the department of Parasitology or Infectious diseases of the LUMC.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Vaccine efficacy | week 12-24, i.e. after challenge
  The protective efficacy of Sm-p80 + GLA-SE to male Sm cercariae measured by the difference in frequency of serum CAA positivity (≥1.0 pg/mL) between the vaccine group and placebo

SECONDARY OUTCOMES:
Safety of (repeated) immunisation | week 0-12
  Frequency and severity of adverse events after (repeated) immunisation with Sm-p80 + GLA-SE
Immunogenicity | week 0-24
  Anti-Sm-p80 IgG antibody titres after (repeated) immunisation with Sm-p80 + GLA-SE measured by ELISA

OTHER OUTCOMES:
Time to CAA positivity | week 12-24
  Comparison of time to positive serum CAA test between the vaccine and placebo groups after exposure to male Sm cercariae at week 12
Peak CAA levels | week 12-24
  Comparison of peak serum CAA concentrations between the vaccine and placebo groups after exposure to male Sm cercariae at week 12
Eosinophils | week 12-24
  Comparison of peak eosinophil counts between the vaccine and placebo groups after exposure to male Sm cercariae at week 12
Antibody responses | week 0-24
  Comparison of (glycan) antibody responses directed against Sm antigens between the vaccine and placebo participants as well as between protected and non-protected participants after exposure to male Sm cercariae at week 12 using protein and glycan arrays
Cellular responses | week 0-24
  Comparison of cellular responses directed against Sm antigens between the vaccine and placebo groups after immunisation and after controlled human infection with Sm cercariae, as well as between protected and non-protected participants
In vitro killing | week 0-24
  Enumeration of the ability of Sm-p80-specific antibodies from human subjects to kill schistosome larvae in vitro from sera collected prior to each vaccination
Transcriptomic profile | week 0-24
  Identification, characterization and comparison of gene expression changes as measured using RNA-seq analysis from PBMC between placebo and vaccine groups

CONTACTS AND LOCATIONS:
Overall Officials: Meta Roestenberg, Prof, Principal Investigator — LUMC

IPD SHARING:
Plan to Share IPD: Undecided